CLINICAL TRIAL: NCT07224633
Title: A Clinical In-Use Evaluation to Assess the Tolerability and Efficacy of a Moisturizer on Acne Prone Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenvue Brands LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS2025SK100252
Record Dates: First submitted 2025-11-01; First posted 2025-11-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12-18

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This is a single-center, monadic clinical study. This study is not randomized or blinded. All subjects will be testing the same IP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group: Moisturizer Use (Experimental)
  Interventions: Other: Use of Barrier Building Moisturizer

INTERVENTIONS:
Other: Use of Barrier Building Moisturizer — Subjects will use the facial moisturizer for 4 weeks according to the following: Apply evenly to your face and neck once daily (or twice daily, if desired) after washing your face with your regularly used facial cleanser for the duration of the study. Record all product applications in the daily diary.

SUMMARY:
The objective of this study is to evaluate the tolerance and efficacy of a facial moisturizer in subjects with mild to moderate acne vulgaris over a 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Fitzpatrick Skin Type of I to VI, targeting the following:

   1. Skin types I, II, III, or IV: 60-70% of enrolled subjects
   2. Skin types V or VI: 30-40% of enrolled subjects
2. Has acne as determined by PI and is undergoing current stable, daily treatment of acne for at least one month prior to study initiation.

   a. Treatments may include but are not limited to, either prescription or over-the counter products, such as: Benzoyl Peroxide, Retinoids (Adapalene, Tretinoin, Tazarotene), Topical Antibiotics and oral antibiotics (if used at least 30 days prior to Visit 1), Topical Dapsone, and Epiduo. Note: use of oral isotretinoin (Accutane) is prohibited. Targeting up to 20 subjects currently using a prescription treatment.
3. Willing to continue his/her normal course of treatment (used at least 30 days prior to Visit 1), for their skin condition with no changes during the study.
4. Generally, in good health based on medical history reported by the subject.
5. Able to read, write, speak, and understand English
6. Individuals have signed the ICD including the photo release and Health Insurance Portability and Accountability Act (HIPAA) disclosure
7. Intends to complete the study and is willing and able to follow the subject responsibilities.

Exclusion Criteria:

1. Has severely sensitive skin and/or has known allergies or adverse reactions to common topical skincare products or to ingredients in the IP or has demonstrated a previous hypersensitivity reaction to any of the ingredients in the IP.
2. Has a clinically significant, unstable medical disorder(s)
3. Is unwilling or unable to comply with the requirements of the protocol.
4. Has a history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
5. Has any surgery and/or invasive medical procedure planned during the course of the study.
6. Has started a hormone replacement therapy (HRT) or hormonal birth control less than 3 months prior to Visit 1 or plans on starting, stopping, or changing doses of HRT or hormonal birth control during the study
7. Presents with a pre-existing or dormant facial dermatologic condition that, in the PI or designee's opinion, may confound the study results or otherwise be inappropriate for study participation (e.g., severe acne, acne conglobata, psoriasis, rashes, skin cancer, many and/or severe excoriations, observable suntan, scars, nevi, tattoo, excessive hair, etc.)
8. Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication.
9. Is taking/using medications or a product that would mask an adverse event (AE) or influence the study results, including:

   1. Steroidal drugs within 2 months before Visit 1
   2. Non-steroidal anti-inflammatory drugs within 5 days before Visit 1
   3. Antihistamines within 2 weeks before Visit 1
   4. Oral isotretinoin (Accutane) within 6 months to Visit 1
   5. Anticancer and immunosuppressive treatments/medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, Remicade, Stelara) currently or within 3 months before Visit 1
   6. Radiation currently or within 1 week before Visit 1
10. Has a history of or a concurrent health condition/situation which, in the opinion of the PI may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
11. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS).
12. Is participating in or planning to receive any professional or aesthetic facial spa procedures during the study.
13. Is simultaneously participating in any other product-use study or has participated in any clinical study on the face in the past 4 weeks.
14. Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor.
15. Is self-reported to be pregnant, breastfeeding, or planning to become pregnant during the study or within 30 days of study completion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2025-10-07 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Investigator's assessment of efficacy | Visit 1 (Screening/Baseline: pre-product use), Visit 2 (Week 1) and Visit 3 (Week 4)
  The Investigator or the expert grader observed efficacy parameters like Visual Dryness, Tactile Surface Roughness, Lack of Radiance/Brightness, Global Fine Lines, Overall Appearance of Pores, Overall Skin Appearance, Skin Blotchiness, Uneven Skin Tone, Lack of Skin Clarity using a 10-point ordinal scale (0=none, 1-3 = mild, 4-6 = moderate, 7-9 = severe).
  A decrease in score compared to baseline indicates an improvement in the efficacy parameter.
Acne Quality of Life Index (AQOLI) 3 Domains and Group Total Scores | Visit 1 (Screening/Baseline: pre-product use) and Visit 3 (Week 4)
  Subjects will complete an Acne Quality of Life Index [Acne-QOLI] using a 1 to 7 scale (1 = extremely, 4 = some, 7 = not at all).
  A decrease in scores indicates improvement.
VISIA Imaging | Visit 1 (Screening/Baseline: pre-product use) and Visit 3 (Week 4)
  Full-face digital images will be taken using the site provided VISIA-CR 5 photographic imaging system.
Investigator's assessment of tolerability | Visit 1 (Screening/Baseline: pre-product use),Visit 2(Week 1) and Visit 3 (Week 4)
  The Investigator will perform a clinical evaluation of each subject's neck and facial skin of Erythema, Edema, Dryness/Scaling, Rash/Irritation using a 4-point ordinal scale (0=none; 1=Mild; 2=Moderate; 3=Severe).
  A decrease in score compared to baseline indicates an improvement in the efficacy parameter.
Subjects' assessment of tolerability | Visit 1 (Screening/Baseline: pre-product use), Visit 2 (Week 1), and Visit 3 (Week 4)
  The Investigator will question each subject for the parameters below regarding the subject's neck and facial skin of Burning, Stinging, Tightness/Dry Feeling , Itching , Peeling/Flaking, Overall sensitivity. Assessments will be scored on a 4-point ordinal scale (0=none; 1=Mild; 2=Moderate; 3=Severe).
  A decrease in score compared to baseline indicates an improvement in the efficacy parameter.
Subjective assessment of efficacy Part A | Visit 1 (Screening/Baseline: pre-product use), Visit 2 (Week 1) and Visit 3 (Week 4)
  Self-assessment regarding the current condition (Appearance of redness associated with pimples, Oiliness of skin, Shininess of skin, Dryness of skin, Flakiness of skin, Skin smoothness, Appearance of pores, Redness of skin, Overall appearance of skin) of facial skin using a 1-10 scale.
  A decrease in score indicates an improvement in the efficacy parameter.
Subjective assessment of efficacy Part B | Visit 1 (Post product use), Visit 2 (Week 1) and Visit 3 (Week 4)
  Self-assessment on efficacy at post product use timepoint. Frequency and percentage of all answers for all questions, and a binomial test (sign test) p-value will be provided for applicable questions.
  A higher percentage of favorable responses with a significant p-value indicates positive subject perceptions of the IP.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research Inc. - Fair Lawn, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No